CLINICAL TRIAL: NCT07244887
Title: Randomized, Triple-Blind, Placebo-Controlled Evaluation of the Clinical Efficacy of Topical Dapsone Gel and Its Effects on Sebum, Erythema and Melanine in Patients With Acne Vulgaris
Brief Title: Randomized, Triple-Blind, Placebo-Controlled Trial of Topical Dapsone Gel in Patients With Acne Vulgaris
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Oya Helin Dundar (Other Government)
Collaborators: Istanbul Training and Research Hospital (Other Government); FARMATEK TARIM SANAYİ MÜMESSİLLİK VE TİCARET ANONİM ŞİRKETİ (Unknown)
Responsible Party: Sponsor-Investigator, Oya Helin Dundar, Dermatology Resident Physician, Istanbul Training and Research Hospital
Organization: Istanbul Training and Research Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SBU-IEAH-AV-DAP7P5-RCT-EC210; Medipol-EC-210 (Other: Istanbul Medipol Univ. Non-Interventional Clin. Research EC)
Record Dates: First submitted 2025-09-10; First posted 2025-11-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Acne Vulgaris
Keywords: Dapsone gel; Topical dapsone 7.5%; Vehicle gel; Mexameter; Erythema; Sebum; Sebumeter; Melanin; Global Acne Grading System (GAGS); Acne Quality of Life Index (AQLI); Acne Lesion Count; Papulopustular acne; Comedonal acne
MeSH Terms: conditions — Acne Vulgaris; Erythema | interventions — Dapsone; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapsone 7.5% Gel (Experimental): Dapsone 7.5% topical gel applied once daily to the entire face for 8 weeks.
  Interventions: Drug: Dapsone 7.5 % gel
- Vehicle Gel (Placebo Comparator): Vehicle (placebo) topical gel without dapsone, identical in base and packaging to the active product; applied once daily to the entire face for 8 weeks.
  Interventions: Drug: placebo vehicle gel

INTERVENTIONS:
Drug: Dapsone 7.5 % gel — Topical dapsone 7.5% gel applied once daily to the entire face for 8 weeks; route: topical; identical-appearing tube to placebo. Manufacturer: Farmatek A.Ş.
  Other Names: topical dapsone 7.5% gel; Vulgarex (country-specific brand)
  Arms: Dapsone 7.5% Gel
Drug: placebo vehicle gel — Vehicle gel without dapsone; same base/excipients and packaging as the active product; applied once daily to the entire face for 8 weeks; route: topical. Manufacturer: Farmatek A.Ş.
  Other Names: placebo gel; vehicle gel
  Arms: Vehicle Gel

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled clinical trial is to learn whether topical 7.5% dapsone gel is effective for treating acne vulgaris in adults.

The main questions are:

* Does dapsone gel reduce the number and severity of acne lesions compared with a placebo (vehicle) gel?
* Does dapsone gel improve skin redness (erythema) and pigmentation (melanin) measured with a Mexameter, and reduce skin oiliness (sebum) measured with a Sebumeter?
* Does treatment with dapsone gel improve patients' quality of life?

Researchers will compare once-daily dapsone gel with a look-alike placebo gel (no active ingredient).

What participants will do:

* Apply either dapsone gel or placebo gel once daily for 8 weeks
* Attend clinic visits at baseline (start), week 4, and week 8
* Have acne lesions counted and graded at each visit
* Have erythema and melanin measured with a Mexameter, and sebum measured with a Sebumeter at predefined facial sites (both cheeks and the glabella)
* Complete a quality-of-life questionnaire at baseline and week 8
* Have standardized photographs taken at each visit

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled clinical trial designed to evaluate the clinical efficacy of topical 7.5% dapsone gel in the treatment of acne vulgaris. The study will also investigate effects on skin biophysical parameters using standardized instruments: erythema and melanin with a Mexameter, and sebum production with a Sebumeter.

Two parallel arms will be included: one group will apply 7.5% dapsone gel once daily, and the other will apply a vehicle (placebo) gel identical in appearance and packaging but without the active ingredient. Randomization will be computer-generated, and both investigators and participants will remain blinded to treatment allocation.

Participants will attend clinic visits at baseline (Day 0), Week 4, and Week 8. At each visit, standardized digital photographs will be taken, and lesion counts will be performed. Lesion assessments will include comedonal and papulopustular counts according to Plewig & Kligman, the Global Acne Grading System (GAGS), and the Investigator's Global Assessment (IGA). At each visit, Mexameter readings (erythema and melanin) and Sebumeter readings (sebum) will be obtained at three predefined facial sites (right cheek, left cheek, glabella/forehead) using triplicate measurements after a standardized acclimatization period. The Acne Quality of Life Index will be administered at baseline and Week 8.

Treatment with dapsone or placebo will continue for 8 weeks, after which the study ends for both arms. Following completion at Week 8, participants may initiate standard acne therapies as clinically indicated outside the study.

The primary focus is to determine whether dapsone gel significantly reduces inflammatory lesion counts compared with placebo at Week 8. Secondary evaluations include changes in comedonal lesion counts, acne severity scores (GAGS and IGA), erythema and melanin indices (Mexameter), sebum levels (Sebumeter), and patient-reported quality of life (Acne-QoL). By combining standardized clinical assessments, validated scoring systems, patient-reported outcomes, and objective biophysical measurements, this trial aims to generate robust evidence regarding the effectiveness of topical 7.5% dapsone in acne management.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 50 years with a clinical diagnosis of acne vulgaris.
* No systemic or topical acne treatment within the past 1 month (30 days).
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Systemic retinoid or systemic antibiotic use within the past 6 months.
* Active dermatologic or systemic disease that could interfere with study participation or assessments.
* Known hypersensitivity to dapsone or any component of the study product.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Inflammatory Lesion Count (Papules/Pustules) | Baseline to Week 8 (with interim assessment at Week 4)
  Mean change from baseline in the number of inflammatory facial acne lesions (papules and pustules) per Plewig & Kligman. Blinded dermatologist, standardized facial mapping. Between-group comparison: topical 7.5% dapsone gel vs vehicle/placebo gel.

SECONDARY OUTCOMES:
Change in Comedonal Lesion Count | Baseline to Week 8 (with interim assessment at Week 4)
  Mean change from baseline in non-inflammatory lesions (open/closed comedones) per Plewig & Kligman. Blinded assessment; standardized counting. Between-group comparison.
Change in Global Acne Grading System (GAGS) Total Score | Baseline to Week 8 (interim at Week 4)
  Mean change from baseline in GAGS (Doshi et al.); higher scores indicate more severe acne. Decrease reflects improvement. Between-group comparison.
Change in Erythema Index (Mexameter) | Baseline to Week 8 (interim at Week 4)
  Mean change from baseline in facial erythema (arbitrary units) measured with Mexameter at three predefined sites (right cheek, left cheek, glabella). Triplicate readings after 15-minute acclimatization; no cosmetics within 24 h. Averages used per visit. Between-group comparison.
Change in Melanin Index (Mexameter) | Baseline to Week 8 (interim at Week 4)
  Mean change from baseline in melanin index (arbitrary units) using Mexameter, same sites/procedure as erythema. Between-group comparison.
Change in Sebum Level (Sebumeter) | Baseline to Week 8 (interim at Week 4)
  Mean change from baseline in sebum level (µg/cm²) measured with a Sebumeter at forehead/cheeks. Triplicate per site; values averaged. Participants refrain from washing face or applying skincare/makeup for ≥4-6 h beforehand. Between-group comparison.
Change in Acne-Specific Quality of Life (Acne-QoL) Total Score | Baseline to Week 8
  Mean change from baseline in Acne-QoL total score (validated instrument). Higher scores indicate better quality of life; an increase reflects improvement. Between-group comparison.
Incidence of Local Cutaneous Adverse Events | Baseline to Week 8 (interim at Week 4)
  Number and proportion of participants with treatment-emergent local reactions (e.g., burning/stinging, dryness, scaling, pruritus, erythema/irritation), graded for severity and relatedness.

CONTACTS AND LOCATIONS:
Overall Officials: Oya Helin Dundar, MD, Principal Investigator — Istanbul Training and Research Hospital, Dept. of Dermatology; Vildan Manav, MD, Assoc. Prof., Study Director — Istanbul Training and Research Hospital, Dept. of Dermatology; Ayse Esra Koku Aksu, MD, Prof., Study Chair — Istanbul Training and Research Hospital, Dept. of Dermatology
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)